CLINICAL TRIAL: NCT06993857
Title: Acute Effect of Forearm Neuromuscular Taping on Maximal Grip Strength, Pressure Pain Threshold, and Muscle Oxygenation in Healthy Collegiate Athletes Post-exercise: A Randomized Controlled Trial.
Brief Title: Acute Effect of Forearm Neuromuscular Taping on Pain, Biological and Functional Variables Post-exercise.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Daniel Martín Vera, Clinical Professor, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-155
Record Dates: First submitted 2025-05-08; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: KINESIOTAPING; NEUROMUSCULAR TAPING

STUDY DESIGN:
Intervention Model Description: Participants are divided into four groups: two experimental groups, one placebo group, and one control group. One experimental group receives NMT with proximal-to-distal tension, while the other receives distal-to-proximal tension. The placebo group receives NMT without tension, and the control group receives no NMT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neuromuscular taping with proximal-to-distal tension (Active Comparator): Neuromuscular taping applied over the forearm with proximal-to-distal tension
  Interventions: Other: Neuromuscular taping applied with proximal-to-distal tension
- Neuromuscular taping applied with distal-to-proximal tension (Active Comparator): Neuromuscular taping applied over the forearm with distal-to-proximal tension
  Interventions: Other: Neuromuscular taping applied with distal-to-proximal tension
- Neuromuscular taping applied with no tension (Sham Comparator): Neuromuscular taping applied with no tension over the forearm
  Interventions: Other: Neuromuscular taping applied with no tension
- No Neuromuscular taping application (No Intervention): No intervention done

INTERVENTIONS:
Other: Neuromuscular taping applied with no tension — Neuromuscular taping applied with no tension over the anterior surface of the forearm before performing an exercise protocol to observe immediate changes in pain pressure, muscle oxygenation and grip strength
  Arms: Neuromuscular taping applied with no tension
Other: Neuromuscular taping applied with distal-to-proximal tension — Neuromuscular taping applied with distal-to-proximal tension over the anterior surface of the forearm before performing an exercise protocol to observe immediate changes in pain pressure, muscle oxygenation and grip strength
  Arms: Neuromuscular taping applied with distal-to-proximal tension
Other: Neuromuscular taping applied with proximal-to-distal tension — Neuromuscular taping applied with proximal-to-distal tension over the anterior surface of the forearm before performing an exercise protocol to observe immediate changes in pain pressure, muscle oxygenation and grip strength
  Arms: Neuromuscular taping with proximal-to-distal tension

SUMMARY:
This study aims to evaluate the acute effect of neuromuscular taping applied to the forearm on maximal grip strength, pressure pain threshold, and muscle oxygenation in healthy university athletes after exercise. Using a randomized controlled trial design, the study aims to provide rigorous evidence that will help clarify the potential benefits of Neuromuscular Taping (NMT) in a sports context. The relevance of this research lies in providing useful information for health and sports professionals, facilitating informed decision-making regarding the use of this technique in daily practice. A randomized controlled trial will be conducted, with participants divided into four groups: two experimental groups, one placebo group, and one control group. One experimental group will receive NMT with proximal-to-distal tension, while the other will receive distal-to-proximal tension. The placebo group will receive NMT without tension, and the control group no NMT application.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years.
* Both genders.
* Body mass index between 18.50 and 23.99 kg/m².
* No musculoskeletal disorders in the last 3 months and intact skin on the forearm.
* No neurological or circulatory disease.
* No additional exercise or treatment during the study.
* No induced fatigue before the experiment.
* Physically active individual (defined as performing at least 150-300 minutes of moderate activity or 75-150 minutes of vigorous activity per week for at least 6 months).

Exclusion Criteria:

* Acute soft tissue injury to the upper extremity in the past month.
* Allergy to NMT or similar drugs.
* History of surgical procedures on the upper extremities.
* Functional impairment of vision or vestibular sensation.
* Frequent use of neuromuscular taping on the upper extremities.
* Analgesic intervention for musculoskeletal pain in the past 3 weeks.
* Participation in a physical therapy rehabilitation program in the past 3 months.
* Serious physical injuries that limit the ability to perform these procedures.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Grip strength | Change from Baseline to immediately after the assigned intervention
  Measurement of grip strength in baseline and immediately after the exercise protocol performance while using NMT (prox-to-distal or distal-to-proximal), sham NMT or no NMT over the anterior surface of the forearm

SECONDARY OUTCOMES:
Muscle oxigenation | Change from Baseline to immediately after the assigned intervention
  Measurement of muscle oxygenation in anterior surface of the forearm (flexor carpi radialis longus) baseline and immediately after the exercise protocol performance while using NMT (prox-to-distal or distal-to-proximal), sham NMT or no NMT over the anterior surface of the forearm
Pressure pain threshold | Change from Baseline to immediately after the assigned intervention
  Measurement of pressure pain threshold in anterior surface of the forearm (flexor carpi radialis longus) baseline and immediately after the exercise protocol performance while using NMT (prox-to-distal or distal-to-proximal), sham NMT or no NMT over the anterior surface of the forearm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldmann A, Schmitz R, Erlacher D. Near-infrared spectroscopy-derived muscle oxygen saturation on a 0% to 100% scale: reliability and validity of the Moxy Monitor. J Biomed Opt. 2019 Nov;24(11):1-11. doi: 10.1117/1.JBO.24.11.115001. PMID 31741352
- [Background] Kuzdzal A, Clemente FM, Kawczynski A, Ryszkiel I, Trybulski R. Comparing The Effects of Compression Contrast Therapy and Dry Needling on Muscle Functionality, Pressure Pain Threshold, and Perfusion after Isometric Fatigue in Forearm Muscles of Combat Sports Athletes: A Single-Blind Randomized Controlled Trial. J Sports Sci Med. 2024 Sep 1;23(1):548-558. doi: 10.52082/jssm.2024.548. eCollection 2024 Sep. PMID 39228772
- [Background] Limmer M, Buck S, de Marees M, Roth R. Acute effects of kinesio taping on muscular strength and endurance parameters of the finger flexors in sport climbing: A randomised, controlled crossover trial. Eur J Sport Sci. 2020 May;20(4):427-436. doi: 10.1080/17461391.2019.1633415. Epub 2019 Jun 29. PMID 31258054
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445